CLINICAL TRIAL: NCT03528785
Title: A Phase II Study of Liposomial IrinoTecan (Nal-IRI) With 5-Fluorouracil, Levofolinic Acid and Oxaliplatin in Patients With Resectable Pancreatic Cancer "nITRo Trial
Brief Title: A Study of Nal-IRI With 5-FU, Levofolinic Acid and Oxaliplatin in Patients With Resectable Pancreatic Cancer
Acronym: nITRo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Ricerche Cliniche di Verona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC2017_01
Record Dates: First submitted 2017-11-09; First posted 2018-05-18 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic Adenocarcinoma; Liposomial IrinoTecan; nal-IRI; Resectable pancreatic cancer
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients will receive a treatment scheme of Irinotecan Liposomal Injection [Onivyde], oxaliplatin, Levofolinic Acid and 5-fluorouracil (5 -FU) on Day 1 and Day 15 of each 28 day cycles.
  Interventions: Drug: Irinotecan Liposomal Injection [Onivyde]; oxaliplatin, 5-FU; Levofolinic Acid

INTERVENTIONS:
Drug: Irinotecan Liposomal Injection [Onivyde]; oxaliplatin, 5-FU; Levofolinic Acid — * Oxaliplatin 60 mg/m2 IV in 120 minutes) on Days 1 and 15 of each cycle
  * Irinotecan Liposomal Injection [Onivyde] (60 mg/m2 IV over 90 minutes) on Days 1 and 15 of each cycle
  * Levofolinic acid (200 mg/m2 IV over 30 minutes) on Days 1 and 15 of each cycle
  * 5FU (2.400 mg/m2 IV over 46 hours) on Days 1 and 15 of each cycle

SUMMARY:
Rational:Pancreatic cancer is a systemic disease at the time of diagnosis, even among patients with apparent localized disease. Surgical resection is the only potentially curative therapy for pancreatic cancer, but in patients who undergo surgery and postoperative therapy, metastatic relapse remains common and no more than 20% of patients achieve 5-year survival.

Because of this aggressive biologic behavior, an increasing interest is growing about preoperative treatments in resectable pancreatic cancer.

The combination chemotherapeutic regimen with irinotecan + 5-fluorouracil (5-FU)/leucovorin (LV) + oxaliplatin (FOLFIRINOX) is an effective choice for first line treatment in patients affected by advanced pancreatic cancer, and in this setting it achieved a Disease Control Rate of 70.2 % (10). In this regard, FOLFIRINOX is currently explored as preoperative regimen in a number of clinical trials in resectable pancreatic cancer.

A critical challenge in this field remains the introduction in these combination treatments of the most novel and effective agents such as nalIRI, in order to obtain a more profound tumor shrinkage, to increase the rate of R0 resections, to allow an early treatment of occult micrometastatic disease, and eventually, to improve survival in patients with resectable pancreatic cancer.

This study proposal is designed to address this challenge. Preliminary results, collected during the Part 1 Dose Escalation of a current clinical trial performed in mPDAC, show that dose of nal-IRI: 60 mg/m2, Oxaliplatin: 60 mg/m2, 5-FU/LV: 2400/400 mg/m2 is safe.

DETAILED DESCRIPTION:
This is a study to determine the proportion of patients affected by resectable pancreatic cancer who achieve R0 resection after a perioperative 6-cycle chemotherapy, 3 pre- and 3 post-surgery, in the absence of disease progression or unacceptable toxicity.

All patients in the program will be identified by a unique identifier number assigned sequentially.

Patients will receive a treatment scheme of nal-IRI, oxaliplatin, Levofolinic Acid and 5-fluorouracil (5 -FU) on Day 1 and Day 15 of each 28 day cycles.

C1D1 is a fixed day, C1D15 and Day 1 and Day 15 of all subsequent cycles should be performed with a window of ± 2 days.

Patients achieving stable disease or better will undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients will receive an additional 3 cycles of nal-IRI, oxaliplatin, Levofolinic Acid and 5-fluorouracil (5 -FU) treatment in the absence of disease progression or unacceptable toxicity.

Tumor responses will be assessed after 3 cycles of preoperative treatment and after 3 cycles of postoperative treatment or sooner if the treating physician suspects disease progression based on clinical signs and symptoms. All treatment decisions will be based on the local radiologist and/or treating physician assessment of disease status.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide written informed consent.
2. ≥ 18 years of age.
3. Histologically or cytologically confirmed adenocarcinoma of exocrine pancreas.
4. Patients must have measurable disease in the pancreas, with no evidence of metastatic disease on imaging of the chest, abdomen and pelvis (contrast-enhanced CT or MRI abdomen with contrast instead of abdominal CT); PET scans alone will not be adequate alternatives.
5. The primary tumor must be surgically resectable, defined as:

   1. no involvement (abutment or encasement) of the major arteries (celiac, common hepatic and/or superior mesenteric artery);
   2. no involvement or <180° interface between tumor and vessel wall of the portal vein, superior mesenteric vein and/or portal vein/splenic vein confluence.
6. Adequate hepatic, renal and hematological function.

Exclusion Criteria:

1. Serum total bilirubin ≥2 x ULN (biliary drainage is allowed for biliary obstruction).
2. Severe renal impairment (CLcr ≤ 30 ml/min).
3. Inadequate bone marrow reserves as evidenced by:
4. ANC ≤ 1,500 cells/μl; or Platelet count ≤ 100,000 cells/μl; or Hemoglobin ≤ 9 g/dL
5. KPS < 60
6. Patients who received previous chemotherapy or radiotherapy for pancreatic disease.
7. Any clinically significant disorder impacting the risk-benefit balance negatively per physician's judgment.
8. Any clinically significant gastrointestinal disorder, including hepatic disorders, bleeding, inflammation, occlusion, or diarrhea > grade 2.
9. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) in last 6 months.
10. NYHA Class III or IV congestive heart failure, ventricular

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients achieving R0 resection after preoperative nanoliposomal irinotecan (nal-IRI), Oxaliplatin, Leucovorin (LV), 5-FluoroUracil (5-FU) | 4-8 weeks after the completion of 3 courses of treatment
  Number of patients achieving R0 resection after preoperative nanoliposomal irinotecan (nal-IRI), Oxaliplatin, Leucovorin (LV), 5-FluoroUracil (5-FU)

SECONDARY OUTCOMES:
To determine 2-year overall survival (OS) | 2 years
  (OS)
determine disease-free survival (DFS) | through study completion, an average of 2 years
  (DFS)
estimate frequency and severity of adverse events associated with chemotherapy | through study completion, an average of 2 years
  AE
determine overall response rate (ORR) following preoperative chemotherapy | through study completion, an average of 2 years
  ORR
estimate proportion of patients going to surgery for resection after preoperative chemotherapy | through study completion, an average of 2 years
  estimate proportion of patients going to surgery for resection after preoperative chemotherapy
estimate pathologic response rate (pCR) | through study completion, an average of 2 years
  (pCR)
assess lymph node status | through study completion, an average of 2 years
  assess lymph node status
assess surgical mortality | through study completion, an average of 2 years
  assess surgical mortality
assess surgical morbidity | through study completion, an average of 2 years
  assess surgical morbidity

CONTACTS AND LOCATIONS:
Overall Officials: stefano milleri, Dr, Study Director — centro ricerche cliniche
Locations (1):
- Centro Ricerche Cliniche, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPDs published
Supporting Information: Study Protocol, CSR
Time Frame: starting 6 months after publication

REFERENCES:
- [Derived] Simionato F, Zecchetto C, Merz V, Cavaliere A, Casalino S, Gaule M, D'Onofrio M, Malleo G, Landoni L, Esposito A, Marchegiani G, Casetti L, Tuveri M, Paiella S, Scopelliti F, Giardino A, Frigerio I, Regi P, Capelli P, Gobbo S, Gabbrielli A, Bernardoni L, Fedele V, Rossi I, Piazzola C, Giacomazzi S, Pasquato M, Gianfortone M, Milleri S, Milella M, Butturini G, Salvia R, Bassi C, Melisi D. A phase II study of liposomal irinotecan with 5-fluorouracil, leucovorin and oxaliplatin in patients with resectable pancreatic cancer: the nITRO trial. Ther Adv Med Oncol. 2020 Sep 4;12:1758835920947969. doi: 10.1177/1758835920947969. eCollection 2020. PMID 33403007